CLINICAL TRIAL: NCT01010373
Title: Application of AS101 in Combination With Chemotherapy for Elderly Acute Myeloid Leukemia (AML) and Myelodysplastic Syndrome (MDS)
Brief Title: Safety and Efficacy Study of AS101 to Treat Elderly Acute Myeloid Leukemia (AML) and Myelodysplastic Syndrome (MDS) Patients
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: The sponsor is currently focusing on different indications
Sponsor: BioMAS Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #77REV00
Record Dates: First submitted 2009-11-09; First posted 2009-11-10 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome
Keywords: Primary Acute Myeloid Leukemia (AML) and Myelodysplastic Syndrome (MDS) induced AML.
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — ammonium trichloro(dioxoethylene-O,O'-)tellurate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AS101 infusions (Experimental): In addition to induction chemotherapy AS101 will be given intravenously. The patient will also receive AS101 infusions during the time break till the next chemotherapy course, as long as the patient does not achieve complete remission and the platelet count is <20,000/μl; ANC <1000. AS101 will be administered likewise up to two consolidation or equivalent chemotherapy courses (re-induction or salvage in the event that no CR is achieved following first induction chemotherapy), i.e., total of three chemotherapy courses.
  Interventions: Drug: AS101

INTERVENTIONS:
Drug: AS101 — 3 mg/m2 AS101 will be given intravenously (IV) three times per week.

SUMMARY:
The purpose of this study is to determine whether addition of AS101 to the standard chemotherapy regimen is effective in the treatment of newly diagnosed elderly (≥60) AML patients and AML transformed myelodysplastic syndrome (MDS) patients.

DETAILED DESCRIPTION:
AML patients frequently develop cytopenia, which can result in life-threatening bleeding and infections. Despite the administration of prophylactic platelet transfusions, these patients remain at risk of clinically significant hemorrhage. There is a growing need for new, innovative strategies, because the outcome for AML patients, particularly for the older ones, has not substantially changed in the last three decades. Thus, novel compounds to target the tumor cell's resistance to chemotherapeutic agents are essential for the improvement of patients' prognoses. AS101 is a non-toxic, organic, tellurium-based small compound with immunomodulating properties which have previously shown bone marrow sparing effect. In addition in preclinical studies AS101 has shown synergistic effect with several cytotoxic drugs. This study will investigate the safety and efficacy of AS101 formulation in combination with the standard therapy for newly diagnosed elderly AML and AML transformed MDS patients.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of primary AML or AML transformed myelodysplastic syndrome (MDS) with FAB classification other than M3 as proven by bone marrow aspiration.
* Age ≥60 years.
* ECOG performance status of 0-2 (Karnofsky >60%).
* Adequate renal functions: Serum Creatinine < 2 times the upper limit of normal (ULN).
* Adequate hepatic function: serum AST and ALT ≤ 3 x ULN.
* Patients with reproductive potential must use an effective contraceptive method through the study. Patients must receive contraceptive and/or fertility counseling prior to entering the study, i.e., information on sperm banking, etc.

Exclusion Criteria:

* Patients receiving any other investigational agents.
* Symptomatic CNS involvement.
* History of pancreatitis or active alcohol abuse.
* Histologic diagnosis of FAB M3 AML.
* Life expectancy of less than 1 month.
* Patient receives Myelotarg (ozogamicin gemtuzumab).
* Use of hematopoietic growth factors such as G-CSF within 1 week prior to treatment initiation.
* Pregnant or lactating females.
* Patient has known human immunodeficiency virus (HIV) infection or known HIV-related malignancy; Patient has active hepatitis A, B or C infection.
* Active, uncontrolled, systemic infection considered opportunistic, life threatening, or of clinical significance at the time of treatment, or any severe concurrent disease which, in the opinion of the investigator, would make the patient inappropriate for trial entry.
* The patient has had congestive heart failure - New York Heart Association (CHF-NYHA) grade II or higher, and/or myocardial infarction within the last 12 months, or any cardiac disorder which, in the opinion of the Investigator, could put the patient at risk of clinically relevant arrhythmia.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Time (days) to reach platelet counts ≥20,000/µl after first induction course and post-remission chemotherapy courses. | Continously during study and maximum 6 months from the beginning of the study.

SECONDARY OUTCOMES:
To assess safety and tolerability of AS101. | Continously during study and maximum 6 months from the beginning of the study.
Reduction in bone marrow blasts from baseline throughout the study period. | Continously during study and maximum 6 months from the beginning of the study.
Time (days) to reach platelets counts ≥50,000/µl after first induction course and subsequent post-remission chemotherapy courses. | Continously during study and maximum 6 months from the beginning of the study.
Time (days) to reach platelets counts ≥100,000/µl after first induction course and subsequent post-remission chemotherapy courses. | Continously during study and maximum 6 months from the beginning of the study.
Time (days) to reach the maximum platelets counts after chemotherapy courses throughout the study period. | Continously during study and maximum 6 months from the beginning of the study.
To evaluate the number of platelet transfusions through the study period. | Continously during study and maximum 6 months from the beginning of the study.
To measure the incidence and severity of bleeding events using the World Health Organization (WHO) Bleeding Scale, during the treatment and follow-up periods. | Continously during study and maximum 6 months from the beginning of the study.
To assess a correlation between VLA-4 expressions level of leukemia blasts in vitro and the response to treatment in terms of blasts percent. | Continously during study and maximum 6 months from the beginning of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel